CLINICAL TRIAL: NCT00003572
Title: Non-Myeloablative Allogeneic Bone Marrow Transplant for Hematologic Malignancies
Brief Title: Total-Body Irradiation, Tacrolimus, and Mycophenolate Mofetil Plus Bone Marrow Transplantation in Treating Patients With Hematologic Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066639, J9845; R01CA067782 (NIH); P30CA006973 (NIH); JHOC-98070603; JHOC-9845; NCI-H98-0023
Record Dates: First submitted 1999-11-01; First posted 2004-02-20 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; Waldenstrom macroglobulinemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; chronic phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Hodgkin Disease; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic-Phase; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Mycophenolic Acid; Tacrolimus; Radiotherapy

INTERVENTIONS:
Biological: peripheral blood lymphocyte therapy
Drug: mycophenolate mofetil
Drug: tacrolimus
Procedure: allogeneic bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Bone marrow transplantation may be able to replace immune cells that have been destroyed by radiation therapy used to kill tumor cells. Sometimes the transplanted cells can make an immune response against the body's normal tissues. Mycophenolate mofetil and tacrolimus may be an effective treatment for graft-versus-host disease caused by bone marrow transplantation.

PURPOSE: Phase II trial to study the effectiveness of total-body irradiation, tacrolimus, and mycophenolate mofetil plus bone marrow transplantation in treating patients with hematologic cancers.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether sustained engraftment of HLA identical sibling marrow can be achieved in patients treated with total body irradiation before transplant and tacrolimus and mycophenolate mofetil after transplant. II. Document the nonhematologic toxicities of this regimen. III. Characterize immune reconstitution of patients during this treatment regimen. IV. Document the incidence of aplasia and graft-versus-host disease associated with donor leukocyte infusions when administered after this regimen.

OUTLINE: Patients receive total body irradiation in a single fraction on day -1. Tacrolimus is given orally twice per day on days -1 to 50. Mycophenolate mofetil is given orally on day 0 and twice per day on days 1 to 28. Patients receive donor bone marrow infusion on day 0. Patients are evaluated on days 56, 180, 292, and 365. If there is donor engraftment, donor chimerism is less than 80%, there is no active graft-versus-host disease, no disease progression, less than 50% decrease in donor cell chimerism from last measurement, and the patient is not taking immunosuppressive agents, then donor leukocyte infusions are administered on days 70, 194, and 306. Patients are followed annually for 5 years.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Must have a 6 antigen HLA identical related donor and one of the following diseases: -Acute myelogenous leukemia in high risk first complete remission or second or greater complete remission -Acute lymphocytic leukemia in high risk first complete remission or second or greater remission -Chronic myelogenous leukemia in chronic phase -Indolent non-Hodgkin's lymphoma (NHL) or aggressive NHL in complete or partial remission, not eligible for autologous bone marrow transplant (ABMT) -Multiple myeloma in complete or partial response -Myelodysplastic syndrome -Stage III or IV chronic lymphocytic leukemia -Hodgkin's disease after first complete remission Patients must also have one of the following high risk features: -Age 55-70 -Age 18-54 must have one of the following conditions: LVEF 35-44% FEV1 or FVC 40-49% Bilirubin 2.1-3.0 mg/dL, AST 71-175, or ALT 81-200 Creatinine 2.1-3.0 mg/dL Disease recurrence less than 1 year after ABMT Between 18 to 24 months of prior chemotherapy (12 to 24 months for multiple myeloma)

PATIENT CHARACTERISTICS: Age: 18 to 70 Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin less than 3.1 mg/dL Renal: Creatinine less than 3.1 mg/dL Cardiovascular: LVEF at least 35% Pulmonary: FEV1 and FVC at least 40% of predicted (60% for patients who have received thoracic or mantle radiotherapy) Other: Not pregnant Fertile patients must use effective contraception Not HIV positive

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1998-08; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ephraim J. Fuchs, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins Oncology Center, Baltimore, Maryland, United States